CLINICAL TRIAL: NCT02892669
Title: Predictive Value of Heart Rate Variability on Outcome in Patients Admitted to the Intensive Care Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: RRV ICU ADMISSION
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients admitted to the intensive care department
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study — non interventional study

SUMMARY:
This study is designed to evaluate the predictive value of heart rate variability on medial outcome in patients admitted to the intensive care department

ELIGIBILITY:
Inclusion Criteria:

* adults admitted to ICU

Exclusion Criteria:

* rhythm other then sinus
* presence of cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care department
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months

SECONDARY OUTCOMES:
ICU stay | 6 months
Hospital stay | 6 months

IPD SHARING:
Plan to Share IPD: No